CLINICAL TRIAL: NCT02654171
Title: A Randomized, Double-blind, Placebo-controlled, 2-Part Study of Orally Administered AK0529 to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Effect of Single and Multiple Dosing in Hospitalized Infants With Respiratory Syncytial Virus Infection
Brief Title: Viral Inhibition in Children for Treatment of RSV
Acronym: VICTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Ark Biosciences Pty Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK0529-1003
Record Dates: First submitted 2016-01-04; First posted 2016-01-13 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: RESPIRATORY SYNCYTIAL VIRUS INFECTIONS
Keywords: RSV; AK0529
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AK0529 (Experimental): Subjects will receive single or multiple doses of AK0529 at different dose levels within different cohorts.
  Interventions: Drug: AK0529
- Placebo (Placebo Comparator): Patients who are randomized to the control arm within each cohort will receive the corresponding placebo to AK0529.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0529 — AK0529 is a novel compound being developed for the treatment of RSV infection. The enteric coated drug pellets with sugar core can be administered orally with apple sauce/purée or yoghurt, or by flushing with 10% dextrose water via a nasogastric or other feeding tube, or upon a glucose wafer.
  Arms: AK0529
Drug: Placebo — The placebo was made with the same smell and appearance as AK0529 but without the active ingredients. The placebo supplements are composed primarily of microcrystaline cellulose pellet.
  Arms: Placebo

SUMMARY:
VICTOR is a randomized, double-blind, placebo-controlled, multicenter, 2-part study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antiviral effect of single and multiple dosing of AK0529 in infants hospitalized with RSV infection.

DETAILED DESCRIPTION:
Globally, Respiratory Syncytial Virus (RSV) is recognized as the leading cause of respiratory tract infections in infants and young children and a major cause of hospitalization due to severe respiratory infection. Despite four decades of effort, there are still no effective methods to control RSV infection. Treatment of RSV has been limited to supportive measures. There is an urgent need for safe and effective drugs to treat and prevent RSV disease.

AK0529 is an investigational antiviral agent that targets the RSV fusion protein on the surface of the viral envelope and exerts antiviral activity against RSV by inhibiting viral entry into host cells and preventing fusion protein induced cell-cell fusion. AK0529 was generally well tolerated in healthy volunteers.

This study is designed as a randomized, double-blind, placebo-controlled, multicenter, phase 2 study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antiviral effect of single and multiple dosing of AK0529 in infants hospitalized with RSV infection. It will consist of two parts, Part 1 and Part 2. Each part will consist of three phases, a pre-treatment phase, a treatment phase and post-treatment follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any race or ethnicity with an age adjusted for any prematurity of ≥1 month and ≤24 months.
* Diagnosis of RSV infection by virological means, which may include rapid diagnostic point-of-care testing, within 96 hours preceding screening for Part 1 and 72 hours for Part 2.
* Patient must weigh >3 kg at screening and be within the 10th and 90th percentiles (inclusive) for the patient's age, based on the local child growth standards, i.e. the Australian Paediatric Endocrine Group Growth Charts.
* The parent / legal guardian of the patient must have provided written informed consent for the patient to participate.
* For patients aged <12 months, an occipito-frontal head circumference within the normal range for age and gender.

Exclusion Criteria:

* The patient has taken, is currently taking or requires any restricted medications.
* Patient is known to be HIV-positive (or the mother, if the potential patient is a child aged <6 months).
* Participation in an investigational drug or device study within 30 days prior to the date of screening.
* Requires vasopressors or inotropic support at the time of enrolment.
* Concurrent gastrointestinal conditions that could, in the opinion of the investigator, prejudice absorption of the Investigational Medicinal Product (e.g. protracted vomiting, malabsorption syndrome, a history of necrotising enterocolitis with consequent short gut syndrome).
* Bronchopulmonary dysplasia or chronic lung disease requiring assisted ventilation at the time of enrolment.
* Diminished ventilatory reserve at risk for hypercapnia (e.g. pulmonary hypoplasia, sequestration syndromes, cystadenomatoid malformation, a history of surgery for diaphragmatic hernia).
* Left to right shunt meriting corrective therapy.
* Renal failure including renal anomalies likely to be associated with renal insufficiency (e.g. clinical conditions of renal dysplasia, polycystic renal disease, renal agenesis).
* Clinical evidence of hepatic decompensation (e.g. hepatic disorder with associated coagulopathy or associated encephalopathy).
* Cerebral palsy with microcephaly, chronic or persistent feeding difficulties or seizures.
* Symptomatic because of inborn errors of metabolism (e.g. mitochondrial disorders, disorders of carbohydrate metabolism, glycogen storage disorders).
* Congenital or acquired immunodeficiency (e.g. congenital agammaglobulinaemia, common variable immunodeficiency, immunosuppressive therapy other than glucocorticoid or montelukast therapy forming part of care directed by the treating physician).
* For Part 2 of this study, children with a history of having received palivizumab or any other monoclonal agent directed against RSV in the preceding 120 days. This exclusion criterion does not apply to Part 1.
* Evidence of active or uncontrolled respiratory, cardiac, hepatic, central nervous system or renal disease unrelated to RSV infection at baseline or any other medical condition that in the opinion of the investigator renders the patient unsuitable for enrolment.
* A history of epilepsy or seizures including febrile seizures.
* Allergy to test medication or constituents.
* Weight less than 10th percentile or greater than 90th percentile for age and gender adjusted for any prematurity.
* The patient's parent or legally acceptable representative is an employee of the investigator or the study center, with direct involvement in the proposed study or other studies under the direction of that investigator of the study center, or any family members of the employees or the investigator.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events during the study | Day -4 to single dose Day 7 (Part 1) and Day -3 to multiple dose Day 14 (Part 2)
Subject withdrawals due to Adverse Events | Day -4 to single dose Day 7 (Part 1) and Day -3 to multiple dose Day 14 (Part 2)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to infinity (AUC) | Pharmacokinetic samples will be taken predose, 2, 4, 6, 12, 18, 24 hours postdose on Day 1, 48 hours postdose (Part 1 and Part 2) and Day 5 (Part 2 )
  For patients without intravenous cannulation, samples will be collected at pre-dose, 2, 6 and 12 hours post-dose on Day 1.
Maximum plasma concentration of AK0529 (Cmax) | Pharmacokinetic samples will be taken predose, 2, 4, 6, 12, 18, 24 hours postdose on Day 1, 48 hours postdose (Part 1 and Part 2) and Day 5 (Part 2 )
  For patients without intravenous cannulation, samples will be collected at pre-dose, 2, 6 and 12 hours post-dose on Day 1.
Plasma concentration of AK0529 at 12 hours postdose (C12) | Pharmacokinetic samples will be taken predose, 2, 4, 6, 12, 18, 24 hours postdose on Day 1, 48 hours postdose (Part 1 and Part 2) and Day 5 (Part 2 )
  For patients without intravenous cannulation, samples will be collected at pre-dose, 2, 6 and 12 hours post-dose on Day 1.
Apparent total body clearance (CL/F) | Pharmacokinetic samples will be taken predose, 2, 4, 6, 12, 18, 24 hours postdose on Day 1, 48 hours postdose (Part 1 and Part 2) and Day 5 (Part 2 )
  For patients without intravenous cannulation, samples will be collected at pre-dose, 2, 6 and 12 hours post-dose on Day 1.
Apparent central compartment volume of distribution (Vc/F) | Pharmacokinetic samples will be taken predose, 2, 4, 6, 12, 18, 24 hours postdose on Day 1, 48 hours postdose (Part 1 and Part 2) and Day 5 (Part 2 )
  For patients without intravenous cannulation, samples will be collected at pre-dose, 2, 6 and 12 hours post-dose on Day 1.
Area under curve change of viral load | From baseline to Day 5
  The antiviral effects in infants hospitalized with RSV are to be determined by measuring the RSV viral load area under the curve in nasal, pharyngeal and tracheal washes / aspirates from baseline to last administration of study medication (Day 5).
Incidence of F-protein genotypes | Specimen will be collected predose and 24 hours postdose on Day 1 (Part 1) and on Day 1-5 (Part 2).
  The incidence of F-protein genotypes associated with reduced sensitivity to IMP will be evaluated.
Change of symptom score | From baseline to Day 1 (Part 1) and up to Day 5 after multiple drug administration (Part 2).
  To evaluate the change of RSV related symptom score in AK0529 arms compared with the change in placebo arm after treatment. The total score is reported with a range from 0 to 12. A decreasing value of total score represents clinical improvement. Subscales are not applicable in this symptom score.

CONTACTS AND LOCATIONS:
Overall Officials: Ark Clinical Trial, Study Director — info@arkbiosciences.com
Locations (28):
- Australia (3):
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Lady Cilento Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
- Prince of Wales Hospital, Shatin, Hong Kong
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Ruth Rappaport Children's Hospital, Haifa
  - Schneider Children's Medical Center, Petach Tikvah
- Lebanon (4):
  - American University of Beirut Medical Center, Beirut
  - Makassed General Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Saint George Hospital University Medical Center, Beirut
- Malaysia (5):
  - Hospital Tuanku Jaafar, Seremban, Negeri Sembilan
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Selayang, Batu Caves, Selangor
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - University Malaya Medical Center, Kuala Lumpur
- Poland (3):
  - Specjalistyczny Zespół Opieki Zdrowotnej nad Matką i Dzieckiem w Poznaniu, Poznan, Greater Poland Voivodeship
  - Nowy Szpital w Świeciu, Gmina Świecie, Kujawy-Pomerania
  - Szpital im. Świętej Jadwigi Śląskiej w Trzebnicy, Trzebnica, Trzebnica County
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (4):
  - Cukurova University Balcali Hospital, Adana, Adana
  - Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Eskişehir
  - Ege University Medical Faculty, Izmir, İzmir
  - Marmara University Faculty of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Result] Huang LM, Schibler A, Huang YC, Tai A, Chi H, Chieng CH, Wang JL, Goldbart A, Tang SP, Huang YC, George S, Alabaz D, Bentur L, Su SC, de Bruyne J, Karadag B, Gu F, Zou G, Toovey S, DeVincenzo JP, Wu JZ. Safety and efficacy of AK0529 in respiratory syncytial virus-infected infant patients: A phase 2 proof-of-concept trial. Influenza Other Respir Viruses. 2023 Jul 25;17(7):e13176. doi: 10.1111/irv.13176. eCollection 2023 Jul. PMID 37502622